CLINICAL TRIAL: NCT00262808
Title: A PHASE II Study of GM-CSF As Pre- And Post-operative Adjuvant Therapy For Stage II And III Colon Cancer
Brief Title: GM-CSF and Combination Chemotherapy in Treating Patients Who Are Undergoing Surgery for Stage II or Stage III Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000448633; URCC-U1203; URCC-RSRB-09956; BRLX-001-0837; DUMC-7135-05-5R0
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — sargramostim; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: sargramostim
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy or kill tumor cells. Drugs used in chemotherapy, such as fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving combination chemotherapy after surgery may kill any remaining tumor cells. Sometimes, after surgery, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient.

PURPOSE: This phase II trial is studying how well GM-CSF and combination chemotherapy work in treating patients who are undergoing surgery for stage II or stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of neoadjuvant and adjuvant sargramostim (GM-CSF) and adjuvant chemotherapy in patients with resectable stage II or III colon cancer.
* Determine the efficacy, in terms of enhanced tumor-associated macrophage response, of this regimen in these patients.

Secondary

* Determine overall survival and time to progression in patients treated with this regimen.

OUTLINE:

* Neoadjuvant therapy and surgery: Patients receive sargramostim (GM-CSF) subcutaneously (SC) once daily beginning between days -16 and -12 and continuing until day -1. Patients undergo surgical resection on day 0. Patients with stage I or IV disease are removed from the study. All other patients proceed to adjuvant chemotherapy or observation.
* Adjuvant chemotherapy or observation: Patients with high-risk stage II or any stage III disease are assigned to group 1 or 2. Patients with low-risk stage II disease are assigned to group 3.

  * Group 1 (adjuvant therapy for high-risk stage II disease): Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV on days 1, 8, 15, 22, 29 and 36. Patients also receive GM-CSF SC once daily on days 50-54. Treatment repeats every 56 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Group 2 (adjuvant therapy for stage III disease): Patients receive adjuvant chemotherapy and GM-CSF as in group 1. Alternatively, patients may receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. These patients also receive GM-CSF SC once daily on days 10-14 of every fourth course. Treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * Group 3 (low-risk stage II disease): Patients undergo observation only every 3 months.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon

  * Stage II or III disease
  * No carcinoma in situ
  * No perforated or obstructed tumors
  * No dual primary lesions by colonoscopy or barium enema
* Resectable disease

  * Distal and proximal bowel end must be > 5 cm from tumor
  * Tumor must not extend below peritoneal reflection
* No distant intra-abdominal metastases (even if resected)
* No rectal cancer

  * No tumors that require opening of the pelvic peritoneum to define the extent of disease

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia

Immunologic

* No ongoing or active infection
* No allergy to yeast or yeast-based products
* No allergy to sargramostim (GM-CSF)
* No allergy to fluorouracil
* No allergy to leucovorin calcium

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of Crohn's disease
* No history of ulcerative colitis
* No other malignancy within the past 3 years except superficial squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy, including fluorouracil, for colon cancer
* No other concurrent chemotherapy

Radiotherapy

* No prior radiotherapy for colon cancer
* No concurrent radiotherapy

Other

* No other prior therapy for colon cancer
* No concurrent immunosuppressant therapy
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a change in tumor-associated macrophage VEGF expression

SECONDARY OUTCOMES:
Disease-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Alok A. Khorana, MD, Principal Investigator — James P. Wilmot Cancer Center
Locations (2):
- United States (2):
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- [Derived] Bourigault P, Skwarski M, Macpherson RE, Higgins GS, McGowan DR. Investigation of atovaquone-induced spatial changes in tumour hypoxia assessed by hypoxia PET/CT in non-small cell lung cancer patients. EJNMMI Res. 2021 Dec 29;11(1):130. doi: 10.1186/s13550-021-00871-x. PMID 34964932